CLINICAL TRIAL: NCT00617435
Title: Impact of Trans Fatty Acids From Natural and Industrial Origin in the Induction of Insulin Resistance Development
Acronym: Trans-Insulin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2006-A00397-44; AU679; 2006-0132
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2009-03

CONDITIONS: Insulin Resistance; Obesity
Keywords: Trans fatty acid; Insulin resistance; Skeletal muscle; Adipose tissue
MeSH Terms: conditions — Insulin Resistance; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- V (Experimental)
  Interventions: Dietary Supplement: vaccenic acid enriched diet
- N (Experimental)
  Interventions: Dietary Supplement: Elaidic acid enriched diet
- J (Experimental)
  Interventions: Dietary Supplement: control diet

INTERVENTIONS:
Dietary Supplement: vaccenic acid enriched diet — The experimental milk fat, entitled "vaccenic acid enriched milk fat" (VAMF), has been obtained by feeding cows with a diet containing sunflower oil.
  Arms: V
Dietary Supplement: Elaidic acid enriched diet — Mixture of vegetable oils (including partially hydrogenated oils)
  Arms: N
Dietary Supplement: control diet — Mixed of different oil
  Arms: J

SUMMARY:
The investigators' project has as for principal objective to understand the impact of trans fatty acids from dairy products and industrial origin on the development of insulin resistance in obese woman. Because of the different isomeric position of the double bound those trans fatty acids may have different metabolic effects.

DETAILED DESCRIPTION:
Women will be included in the study according to their susceptibility to develop a insulin resistance (evaluated starting from the body index of mass IMC superior to 28 kg.m-², of the waist measurement 88 cm). Once included in the study, the volunteers will receive for 4 weeks butter, dairy products and biscuits enriched in stearic, elaidic or vaccenic acid. The volunteers will undergo a measurement of the body composition by biphotonic absorptiometry as well as a complete metabolic assessment (blood and urinary samples, clamp to insulin and biopsies).

ELIGIBILITY:
Inclusion Criteria:

* female
* waist measurement > 88 cm
* body mass index> 28kg/m2
* Affiliated to National Health Insurance
* Subject giving his/her written informed consent
* Subject willing to comply with the study procedures
* Subject considered as normal after clinical examination and medical questionnaire

Exclusion Criteria:

* Reported food allergies
* Currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study
* Hepatic or renal impairments
* Positive serologies to HIV or HCV, determined on blood sample
* pregnant or presently attempting to get pregnant or menopause or lactating Blood donation done less than 2 months before the start of the study
* Chronic pathologies: diabetes, hypertriglyceridemia, hypertension, cardiovascular diseases, chronic inflammatory diseases
* Intestine, cardiovascular, kidney and cancer pathologies in the last 5 years
* Previous heavy intestine surgery (except appendicectomy)
* Previous medical and/or surgery judged by the investigator as incompatible with this study
* High variation (> 5%) of body weight during the last 3 months
* Consuming nutritional supplements which could interfered with lipid metabolism (fish oil capsule, vitamins, soja lecithins,…)
* Heavy consumer of alcohol
* Smoker or ex-smoker who stopped smoking less than 1 month before V0 (more than 5 cigarettes/dy).
* Practising intensive physical exercise (> 5 h per week)
* Vegetarian or vegan
* Being under someone's supervision
* Refusal to be registered on the National Volunteers Data file
* Disliking butter, margarine, cheese, biscuits and/or vegetable oil
* Dietary habits unreliable to controlled food intake
* Being in exclusion on the National Volunteers Data file

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Measure of insulin sensitivity by an hyperinsulinemic- euglycemic clamp. | before and after 4 weeks of diets.

SECONDARY OUTCOMES:
Muscle and adipose tissue biopsies and Body composition | before and after 4 weeks of diet

CONTACTS AND LOCATIONS:
Overall Officials: Yves Boirie, MD, PU-PH, Principal Investigator — UMR1019 INRA - Université Clermont1
Locations (2):
- France (2):
  - Centre de Recherche en Nutrition Humaine Auvergne, Clermont-Ferrand
  - Centre de Recherche en Nutrition Humaine Rhônes-Alpes, Lyon

REFERENCES:
- [Background] Chardigny JM, Malpuech-Brugere C, Dionisi F, Bauman DE, German B, Mensink RP, Combe N, Chaumont P, Barbano DM, Enjalbert F, Bezelgues JB, Cristiani I, Moulin J, Boirie Y, Golay PA, Giuffrida F, Sebedio JL, Destaillats F. Rationale and design of the TRANSFACT project phase I: a study to assess the effect of the two different dietary sources of trans fatty acids on cardiovascular risk factors in humans. Contemp Clin Trials. 2006 Aug;27(4):364-73. doi: 10.1016/j.cct.2006.03.003. Epub 2006 Apr 24. PMID 16632411
- [Derived] Tardy AL, Lambert-Porcheron S, Malpuech-Brugere C, Giraudet C, Rigaudiere JP, Laillet B, Leruyet P, Peyraud JL, Boirie Y, Laville M, Michalski MC, Chardigny JM, Morio B. Dairy and industrial sources of trans fat do not impair peripheral insulin sensitivity in overweight women. Am J Clin Nutr. 2009 Jul;90(1):88-94. doi: 10.3945/ajcn.2009.27515. Epub 2009 May 27. PMID 19474135